CLINICAL TRIAL: NCT05587023
Title: Effect of Ultrasound-guided Left Stellate Ganglion Block on Rapid Recovery of Patients Undergoing Cardiac Valve Replacement and Its Mechanism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhonghua Chen,MD (Other)
Collaborators: Shaoxing Hospital of Zhejiang University (Other)
Responsible Party: Sponsor-Investigator, Zhonghua Chen,MD, Head of anesthesiology, Shaoxing Hospital of Zhejiang University
Organization: Shaoxing Hospital of Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2021-K-Y-294-01
Record Dates: First submitted 2022-10-16; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Left Stellate Ganglion Block Can Quickly Restore the Left Stellate Ganglion; Possible Molecular Mechanism of Left Stellate Ganglion Block
Keywords: ultrasound-guided、 left stellate ganglion block 、on rapid rehabilitation in patients with cardiac Valve replacement

STUDY DESIGN:
Intervention Model Description: Sixty patients with cardiac Valve replacement undergoing cardiopulmonary bypass were randomly divided into experimental group and control group, with 30 patients in each group. All patients signed the informed consent form. Control Group: the control group was injected with 6ml normal saline. Test group: the test group was injected with 0.5% ropivacaine 6ml.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither the experimenters nor the participants knew whether they were taking a Experimental drug or a placebo. To be as objective as possible, the description of the treatment effects and adverse reactions of the subjects, as well as the recording of the various reactions of the experimenters, should be given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): the test group was injected with 0.5% ropivacaine 6ml.
  Interventions: Procedure: stellate ganglion block
- Control group (Placebo Comparator): The control group was injected with 6ml normal saline
  Interventions: Procedure: stellate ganglion block

INTERVENTIONS:
Procedure: stellate ganglion block — The experimental group was given 6ml ropivacaine for stellate ganglion block. In the control group, 6ml saline was used for stellate ganglion block.

SUMMARY:
In this study, Valve replacement patients undergoing cardiopulmonary bypass were randomly divided into control group and experimental group (SGB Group) , main outcome measures: postoperative complications (pulmonary infection, oxygenation injury, arrhythmia, hemorrhage, enteroparalysis, incision infection, renal insufficiency, cognitive impairment, etc.) and 30-day mortality. Secondary outcome measures: Hemodynamics, postoperative extubation time, length of stay and total cost of hospitalization. To investigate the effect of SGB on the rapid recovery of patients with Valve replacement heart disease after cardiopulmonary bypass.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effect of left stellate ganglion block on the incidence and severity of postoperative complications in patients with cardiac Valve replacement undergoing cardiopulmonary bypass, to compare the difference of inflammatory reaction between the control group and the stellate ganglion block group at different time points, and to preliminarily elucidate the molecular mechanism of stellate ganglion block in the protection of cardiac Valve replacement during cardiopulmonary bypass (CPB) . The first part is a prospective study on the effect of left stellate ganglion block on cardiac Valve replacement Hemodynamics during cardiopulmonary bypass (CPB) , the incidence, length of hospital stay, cost of hospital stay, and 30-day mortality of the common Valve replacement complications after cardiopulmonary bypass (pulmonary infection, oxygenation injury, arrhythmia, bleeding, intestinal paralysis, incision infection, renal insufficiency, cognitive impairment, etc.) , to determine the effect of left stellate ganglion block on rapid recovery from cardiac Valve replacement during cardiopulmonary bypass. In the second part, we collected the dynamic changes of inflammatory factors in plasma of control group and patients with stellate ganglion block before and 1,3,6,24 and 72 hours after operation, to explore the molecular mechanisms by which left stellate ganglion block promotes rapid recovery and reduces severe complications in patients with cardiac Valve replacement undergoing cardiopulmonary bypass (CPB) .

ELIGIBILITY:
Inclusion Criteria:

- Sixty patients with cardiac Valve replacement undergoing elective cardiopulmonary bypass, with cardiac function class II-IV and ASAII-IV, aged 18-70 years.

Exclusion Criteria:

- Patients with off-pump cardiac Valve replacement, age > 18 years or > 70 years, cardiac function ≥ III, ASA grade ≥ III, local anesthetic allergy, concomitant immune disease or immunosuppressive status, patients with severe mental disorders who could not cooperate with SGB, abnormal neck anatomy, and failure of stellate ganglion block refused to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | within 1 week after operation
  Pulmonary infection, oxygenation injury, malignant arrhythmia, hemorrhage, enteroparalysis, incision infection, renal insufficiency, cognitive dysfunction and so on

SECONDARY OUTCOMES:
Mortality | Within 30 days after surgery
  Mortality

OTHER OUTCOMES:
The concentration of blood factors in plasma | Within 3 days after surgery
  Plasma levels of IL-6, IL-10 and TNF-α were measured by enzyme-linked immunosorbent assay (Elisa) at 1,3,6,24 and 72 h after operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhonghua Chen,MD, Shaoxing, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No